CLINICAL TRIAL: NCT02975401
Title: Prospective Observational Cohort Study on Robot-assisted Laparoscopic Hernia Repair (rTAPP)
Brief Title: Robotic Utility for Surgical Treatment of Groin Hernias
Acronym: Robust _1
Status: Completed | Type: Observational
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Filip Muysoms, surgeon, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: Robust_1
Record Dates: First submitted 2016-10-24; First posted 2016-11-29 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: rTAPP technique — robot-assisted rTAPP technique
  Other Names: laparoscopic robot-assisted TAPP technique

SUMMARY:
The purpose of this study is the measurement of the evolution of the operation time during the start-up phase of robotic-assisted surgery for the treatment of inguinal hernia's of 50 patients treated in Maria Middelares in laparoscopic rTAPP technique.

DETAILED DESCRIPTION:
Minimally invasive hernia repair by laparoscopy is the standard treatment in adult patients in Maria Middelares, Ghent. A previously conducted study demonstrated that the symptoms of patients with inguinal hernias (verified via EuraHS Quality of Life score) can be effectively treated and the technique has a low recurrence rate and low frequency of long-term side effects.

Robot-assisted laparoscopic surgery has become standard in urology for resection of the prostate carcinoma. In general abdominal surgery, a large group of surgeons are currently working on the introduction of robotic-assisted surgery for resection of colon and rectal cancer in their daily practice. The third generation robot (DaVinci Xi), has extended the applicability of this technology within the field of general surgery.

For the surgical treatment of hernia's and other abdominal wall defects (umbilical or/and incisional hernia's), currently only surgeons in the US have experiences in structured treatment programs.

From September 1, 2016 Maria Middelares hospital will introduce robot-assisted surgery, including the laparoscopic TAPP inguinal hernia repair.

Main obstacles to the introduction of robot technology in abdominal wall surgery are prolonged preparation time in the operating room required for installation of the robot, and higher material costs related to the robot-assisted surgery. However, there are few precise data available on the exact size of extra time or increased costs related to the introduction of robotic assisted surgery in a program for abdominal surgery.

The purpose of this study is the measurement of the evolution of the operation time during the start-up phase of robotic-assisted surgery for the treatment of inguinal hernias by 50 patients in Maria Middelares hospital.

ELIGIBILITY:
Inclusion Criteria:

* 50 patients selected and operated by the PI.

Exclusion Criteria:

* patients under the age of 18
* pregnancy
* BMI > 35
* recurrent groin hernia
* no Informed Consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients who are scheduled for laparoscopic repair of a unilateral or bilateral inguinal hernia. A total of 50 patients will be enrolled in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
duration of the operation | from the start of the operation until the end of the operation, approximately 3 hours
  Recording of the operation time needed for robot-assisted TAPP groin hernia repair

SECONDARY OUTCOMES:
intra-operative complications | until 4 weeks post-operative
  Intra-operative complications registered until 4 weeks post-operative
post-operative complications | until 4 weeks post-operative
  Post-operative complications detected until 4 weeks after hernia repair by clinical follow up.
Quality of Life | until 4 weeks post-operative
  Quality of Life measured with the EuraHS QoL score preoperative and until 4 weeks after hernia repair by clinical follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, MD, PhD, Principal Investigator — Maria Middelares hospital
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muysoms F, Van Cleven S, Kyle-Leinhase I, Ballecer C, Ramaswamy A. Robotic-assisted laparoscopic groin hernia repair: observational case-control study on the operative time during the learning curve. Surg Endosc. 2018 Dec;32(12):4850-4859. doi: 10.1007/s00464-018-6236-7. Epub 2018 May 15. PMID 29766308